CLINICAL TRIAL: NCT04449965
Title: The Efficacy of Topical Povidone-Iodine Rinses in the Management of the Coronavirus Disease 2019 (COVID-19)
Brief Title: Povidone-Iodine Rinses in the Management of COVID-19
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The site struggled with patient recruitment as we were not able to reach patients with COVID-19
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Assistant Clinical Professor, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Betadine COVID-19
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Covid19
Keywords: Povidone - Iodine; Covid19; Self-Isolation
MeSH Terms: conditions — COVID-19 | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator will be blinded to whether or not the patients are receiving either active treatments or placebo, and assignments will be concealed throughout the study. The patients will know if they are in the nasal gel spray or rinse group but will be blinded to whether or not they are receiving the active treatment or placebo if they are randomized into the rinse group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PVP-I sinus rinses and throat gargles (Experimental): Participants will dilute 7 mL of 10% PVP-I into 300 mL of saline for a final concentration of 0.23% available iodine. They will be instructed to rinse each nostril with 120ml (total 240mL) in a NeilMedTM sinus rinse bottle, and gargle with 60 mL of the solution.
  Interventions: Drug: Povidone-iodine
- Placebo sinus rinses and throat gargles (Placebo Comparator): Participants will dilute 7 mL of PVP-I placebo into 300 mL of saline. They will be instructed to rinse each nostril with 120ml (total 240mL) in a NeilMedTM sinus rinse bottle, and gargle with 60 mL of the solution.
  Interventions: Drug: Placebo
- PVP-I gel forming nasal spray (Experimental): 0.6% PVP-I gel forming nasal spray will come prepared and ready for participants to use. They will be instructed to use two sprays to each nostril each time they administer the spray.
  Interventions: Drug: Povidone-iodine

INTERVENTIONS:
Drug: Povidone-iodine — This will be performed twice daily for two weeks.
  Other Names: Betadine
  Arms: PVP-I gel forming nasal spray; PVP-I sinus rinses and throat gargles
Drug: Placebo — This will be performed twice daily for two weeks.
  Arms: Placebo sinus rinses and throat gargles

SUMMARY:
The aim of this study is to determine if Povidone iodine (PVP-I) rinses and throat gargles or a PVP-I gel forming nasal spray compared to a placebo (a treatment that has no physical effect to a person) is an effective treatment for patients diagnosed with COVID-19. These patients have been diagnosed with mild/moderate COVID-19 symptoms and sent home for self-isolation. Patients will be instructed to take either of the two treatments or placebo twice daily for two weeks and have follow up visits 2 and 4 weeks after. The participants will also complete study related procedures such as saliva sample collection, and two questionnaires throughout the study period. The investigators hypothesize that COVID 19 positive participants who use either of the Povidone - Iodine treatment will have a reduction in their viral load, develop a negative oral mucosa sample and improve their clinical symptoms.

DETAILED DESCRIPTION:
The proposed study is a prospective randomized double blinded placebo-controlled study of 6-weeks in duration. Patients who have tested positive and diagnosed with COVID-19 within the previous 72 h and who meet the inclusion and exclusion criteria, will be invited to participate in this study.

This study will be involving non-hospitalized patients who are recovering at home. One arm will use betadine sinonasal rinses and a betadine mouth gargle while another arm will act as a control receiving a placebo (a food coloring agent). A third arm will use a 0.6% PVP-I gel forming nasal spray twice daily. A baseline saliva sample will be collected to assure a positive COVID-19 test and to quantify viral load. Repeat saliva samples will be collected every 2 days for 2 weeks, then at 4 weeks and 6 weeks to quantify test status and quantify viral load reduction. WURSS-44 questionnaires will be completed daily for 2 weeks and then again at 4 weeks and 6 weeks. SNOT-22 questionnaires will be completed at baseline and then again at 2 weeks, 4 weeks, and 6 weeks. The investigators will also monitor for worsening of symptoms and the need for hospitalization for the entire 6 week duration of the study.

Upon enrolment in the study after obtaining positive results for COVID-19, demographic data and clinical data will be obtained by the investigators. Patients will be randomly assigned to one of the study arms delineated above by permuted block randomization

The clinical samples that detect COVID-19 are obtained by collecting a saliva sample prior to rinsing. This will avoid confounding by artificially lowering the viral particles sampled and will minimize any potentially inhibitory effects of the intervention compounds on lab detection. The sample will be put into a sterile collection container and stored in the fridge until it is transported to the laboratory for analysis.

Sample Size

Considering the quick turnover and the rapid doubling time in the number of positive cases and the unprecedented nature of this study's design and treatment, the investigators hope to recruit 20 patients in each study arm as a pilot study around this subject matter. To account for a drop-out rate of 25% the investigators plan to recruit 27 patients in each arm.

Analysis

Primary outcomes

1. Time to a negative/undetectable RT-PCR SARS-CoV-2 saliva sample amongst patients rinsing and gargling with 0.23% PVP-I compared to a placebo group measured during the study treatment daily for 2 weeks and at the 4-week and 6-week mark.

   1.1. A Kaplan-Meier curve and log rank test will be used to compare the time to a negative saliva test from the start of the study between patients receiving PVP-I to those receiving the placebo. A hazard ratio of >1 will favor treatment with PVP-I, calculated with a 95% confidence interval by Cox proportional hazards model.

   1.2. The median time to negative swab in the PVP-I group versus the control will be statistically compared using the unpaired Mann-Whitney U test.

   1.3. The proportion of patients with a negative sample will be compared between the PVP-I group and control group at all times points using the Chi-squared test.

   1.4. A subsequent risk factor analysis will be conducted using the cox proportional hazards model, investigating the independent influence of various host and disease factors on the time to a negative sample during the study period. The following relevant factors included in the multivariable regression were identified a priori upon consultation with experienced clinicians at our center: gender, age, smoking status (yes/no), baseline viral load, known baseline lung comorbidity (yes/no) , duration of symptoms before treatment.
2. SARS-CoV-2 viral load changes in the saliva amongst patients rinsing and gargling with 0.23% PVP-I compared to a placebo group measured during the study treatment daily for 2 weeks and at the 4-week and 6-week mark.

   2.1. Logarithmic viral load levels in the saliva samples will be graphed and compared between the PVP-I and placebo group at all time points using the unpaired Mann-Whitney U test. For complete statistical analysis, a value of 1 log base 10 copies/mL will be assigned to samples with undetectable viral levels.
3. Time to a negative/undetectable SARS-CoV-2 saliva sample as well as SARS-CoV-2 viral load changes amongst patients rinsing and gargling with 0.23% PVP-I compared to the 0.6% PVP-I gel forming nasal spray for 2 weeks and at the 4-week and 6-week mark.

3.1. Similar analysis as per 1.1, 1.2, 1.3 and 2.1 above in primary outcomes.

Secondary outcomes

1. Change in symptom scores between the PVP-I group and placebo group as assessed by the SNOT-22 scores collected at baseline and at the 2-week, 4-week and 6-week mark.

   1.1. SNOT-22 scores will be graphed and compared between baseline and each time point for each group separately using the ANOVA with repeated measures test and Bonferroni post hoc test.

   1.2. The change in SNOT-22 scores between baseline and each time point will be compared between groups using the unpaired Mann-Whitney U test.
2. Change in symptom scores between the PVP-I group and placebo group as assessed by the WURSS-44 scores collected daily from baseline for 2 weeks and at the 4-week and 6-week mark.

   2.1. WURSS-44 scores will be graphed and compared between baseline, the 2 week, 4-week and 6-week marks for each group separately using the ANOVA with repeated measures test and Bonferroni post hoc test.

   2.2. WURSS-44 scores will be graphed and compared between baseline and at all time points using the unpaired Mann-Whitney U test.
3. The need for hospitalization between the PVP-I group and placebo group. 3.1. The Kaplan-Meier technique will also be used to compare the need for hospitalization from the start of the study between both groups.
4. The change in SNOT-22 scores, WURSS-44 scores and the need for hospitalization between patients rinsing and gargling with 0.23% PVP-I compared to the 0.6% PVP-I gel forming nasal spray.

4.1. Similar analysis as per 1.1, 1.2, 2.1, 2.2 and 3.1 above in secondary outcomes.

Descriptive statistics (mean, median, SD) will be used to describe demographic characteristics of the patients. Results will be considered statistically significant with p values < 0.05. All statistical analyzes will be performed using RStudio version 3.4.1 (RStudio, Boston, MA, USA).

Assessment of Safety

Safety Monitoring

Patients who experience signs and symptoms of iodine reaction will be noted and the code will be broken so that a discussion can occur between the research supervisor and the patient regarding the use of the topical iodine.

Patients can contact the office anytime if they notice any of the signs or symptoms of iodine reaction and will be seen by the research supervisor (or designate) within 24 hours.

Adverse Events (AE's)

All expected and unexpected adverse events will be recorded and graded by the research supervisor. Stable chronic conditions, which are present prior to the clinical trial entry and do not worsen, are not considered adverse events and will be accounted for in the patient's medical history.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Patients diagnosed with laboratory-confirmed SARS-CoV-2 and the development of COVID-19 compatible symptoms within the last 72 hours before enrolment
* Do not require hospitalization

Exclusion Criteria:

* Sinonasal tumor
* Hypersensitivity to iodine or betadine
* History of thyroid disorder including thyroid cancer, hyperthyroidism and hypothyroidism
* Use of medications for thyroid disorders including thyroxine and carbimazole
* Current use of topical iodine or betadine for another reason
* Participating in any study with therapies directed at COVID-19 that could influence our results
* Are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 positivity in the saliva | A saliva sample will be taken every 2 days for 2 weeks, and again at 4 and 6 weeks
  A saliva sample will be analyzed to monitor the duration of positivity and when test becomes negative for SARS-CoV-2.
Change in the SAR-CoV-2 viral load in the saliva | A saliva sample will be taken every 2 days for 2 weeks, and again at 4 and 6 weeks
  Quantify the amount of SAR-CoV-2 viral load present in the saliva.

SECONDARY OUTCOMES:
Change in Wisconsin Upper Respiratory Symptom Survey (WURSS-44) | daily for 2 weeks, 4 weeks, and 6 weeks
  This is a 44 question, quality of life survey designed to measure different aspects affected by the common cold.
Change Sino nasal Outcome Test (SNOT-22) | baseline, 2 weeks, 4 weeks, 6 weeks
  That includes 22 questions about symptoms and social/emotional consequences of your nasal disorder.
Change in clinical condition | daily for 2 weeks, 4 weeks, and 6 weeks
  We will record and worsening of clinical condition such as, need for hospitalization/oxygen support.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada